CLINICAL TRIAL: NCT04706754
Title: Pan-Canadian Lung Cancer Observational Study (PALEOS)
Status: Recruiting | Type: Observational
Sponsor: William Osler Health System (Other)
Collaborators: Pulse Infoframe (Industry)
Responsible Party: Principal Investigator, Dr. Parneet Cheema, Principal Investigator, William Osler Health System
Other Study IDs: PALEOS
Record Dates: First submitted 2020-05-20; First posted 2021-01-13 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective: Adults aged 18 years or older having a documented lung cancer diagnosis since 2000.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Participants will complete the survey(s) at the initial visit and every 3 months and/or whenever there is an update in their treatment protocol. Patients may also choose to opt out of the surveys and only consent to primary data collection at the site.

SUMMARY:
A multicenter, ambispective observational study focusing on patients diagnosed with lung cancer in Canada identified after January 1, 2000 inclusive. This data will be combined with that from deceased patients identified.

DETAILED DESCRIPTION:
Lung cancer is no longer considered a single entity. In the real world of lung cancer, it consists of many subgroups that are defined in different ways by different clinicians and researchers. In broad categories, these include sociodemographic, molecular, treatment or biomarker driven subgroups, to name a few. As a result, the single site/centre study of lung cancer is not viable, as no single site/centre has adequate numbers of each subgroup to study by themselves. PALEOS is designed to use the power of a multi-institutional study to evaluate these important questions of natural history, treatment patterns, outcomes as they relate to new diagnostic, new biomarker, new treatments. Real world data will be generated by PALEOS. Thus, there will be broader understanding of how treatments and outcomes that were originally studied in the clinical trials setting would now be translated into the real-world setting. The information from this initiative will result in knowledge translation across disciplines.

Centre/Local Principle investigator and/or Co-investigators or their designee will identify potential patients through physician and hospital medical records, as well as clinic patient lists/databases, hospital pharmacy databases, hospital patient access program lists/databases and hospital pathology databases.

Potential prospective patients will be given a PALEOS Study Information Sheet in clinic or via mail/email, via their circle of care. Study staff will contact the patient by phone, or the patient can contact the study staff if they do not want to participate in the study. The ICF will be made available to the participant if they confirm interest in the study or if they provide verbal consent to participate. The ICF will be provided in person at the clinic or verbally if participant is not able to come to the clinic. The consenting process must be documented clearly in the patient study file by the study staff. The PALEOS Study Information Sheet and ICF will also be sent to referring physicians for patients that are eligible. Patients can opt out of the surveys if they choose to and only consent to data collection. Follow-up contact will be done by the study staff in clinic, by phone, email, or virtually.

After enrollment, Initial/baseline survey of standard demographic information will be collected. Medical records will be reviewed by principal investigator, co-investigator or authorized designee. Data abstraction for each patient's medical history will be performed and entered directly into a secured database with minimal identifiers of the participating patient. Participating patient will be added a study specific unique identifier and that will be used to identify the data. Only the de-identified data will be analyzed to assess patient outcomes and results of treatment, as well as to uncover links between clinical data and pathological and molecular subtypes, where applicable. Study operational documents will be updated regularly (at least annually) and will specify which genetic alterations are current priorities for recruitment. The study will begin with ALK, EGFR, ROS1, ERBB2 (HER2), exon 20 EGFR mutation, MET,BRAF, RET, NTRK and KRAS-G12C patients, with the goal of expanding into other rare molecular alterations as and when they are discovered or become relevant . Patient reported outcomes measure for patients with rare molecular alterations will also be captured and analyzed. Patients will be invited to complete health-related quality of life (HRQoL) surveys in English or French language.

The web-based data capture platform will have a patient portal for capturing patient entered data (PED) including demographic data of patient. Patients clinical data will be both retrospective and prospective that will include previous medical records, lab results and clinical testing.. Certified study site personnel will manage collection and data entry of full medical records with patient consent or with REB approved waiver of consent in the patient clinical data (PCD) portal. Data will be uploaded and stored to a secure server that will be a 21 CFR Part 11, GCP, GDPR, HIPAA, NIST, PHIPA and GDPR compliant online data repository. Pulse Infoframe Inc. (Pulse), London, Ontario, Canada, compliant to all the above regulations, will serve as the study data coordinating Center.

ELIGIBILITY:
Inclusion Criteria:

• Adults aged 18 years or older having a documented lung cancer diagnosis since 2000.

Exclusion Criteria:

• Patients that decline to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 years or older having a documented lung cancer diagnosis since 2000 from across participating sites/cancer centers across Canada.
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2020-04-07 (Actual); Primary Completion 2040-04-07 (Estimated); Study Completion 2045-04-07 (Estimated)

PRIMARY OUTCOMES:
Treatment effectiveness | Patients will be followed for at least 5 years, for a total of 25 years
  * To report on the natural history of multiple subgroups of lung cancer patients (regardless of stage) in Canada, from 2000 onwards, using a combination of retrospective and prospective methods that includes diagnostic, molecular alterations, treatment, and outcomes.
  * To report the real-world treatment patterns of all and specific subgroups of lung cancer patients in Canada, across time (from 2000 onwards), geography.
  * To recruit from centres that are representative of Canadian patients seen in both academic and community cancer settings.
Outcome of Patients | Patients will be followed for at least 5 years, for a total of 25 years
  * To evaluate patient-reported outcomes of different subgroups of lung cancer, through all phases of the disease, from diagnosis through to end-of-life.
  * To understand the incidence, prevalence, and outcomes (efficacy and toxicity), and patterns of locoregional and metastatic spread of different subgroups of lung cancer.
  * To understand the evolution of clinical implementation of new diagnostic tests, new biomarker tests, new treatments (whether it be surgical, medical, radiation or other), including access by healthcare teams and patients, their rates of adoption into clinical practice, and retention of over time.
  * To compare the natural history, stage distribution, treatment outcomes such as treatment effectiveness (composite of disease progression or death) and treatment toxicities (where available) across sub-group of patients with tumors that have been molecularly subtyped and identified to have rare molecular alterations.

CONTACTS AND LOCATIONS:
Overall Officials: Parneet Cheema, MD, Principal Investigator — William Osler Health System; Sara Kuruvilla, MD, Principal Investigator — London Health Science Center
Locations (1):
- Milena (Lynn) Vicente, Brampton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided